CLINICAL TRIAL: NCT02230930
Title: Open-label Crossover Trial to Investigate the Efficacy of Treatments in Apomorphine-induced Skin Reactions
Brief Title: Treatment of Apomorphine-induced Skin Reactions: a Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Delayed inclusion - stopped when 10 patients completed the study
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 46934
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease; Apomorphine-induced Skin Reactions
Keywords: Parkinson's disease; Apomorphine; Infusion; Skin reactions; Subcutaneous nodules; Hydrocortisone; Massage; Dilution
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine; Massage; hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Massage with a spiky ball (Active Comparator): Subjects are instructed to massage the apomorphine-induced skin reactions with a spiky ball 3 times a day for 2 minutes for 14 days.
  Interventions: Device: Massage with a spiky ball
- Hydrocortisone cream 1% (Active Comparator): Subjects are instructed to apply hydrocortisone cream 1% once daily for 14 days.
  Interventions: Drug: Hydrocortisone cream 1%
- Subcutaneous hydrocortisone 10mg (Active Comparator): Subjects are instructed to administer subcutaneous hydrocortisone (Solu-Cortef 10mg) prior to apomorphine via the subcutaneous infusion line which is used for administration of apomorphine, for 14 days.
  Interventions: Drug: Subcutaneous hydrocortisone 10mg
- Apomorphine 0.25% (2.5mg/ml) (Active Comparator): Subjects are instructed to dilute apomorphine 0.5% (5mg/ml) with the same volume of physiologic saline (NaCl 0.9%) to 0.25% (2.5mg/ml). Apomorphine will be infused subcutaneously for 14 days.
  Interventions: Drug: Apomorphine 0.25% (2.5mg/ml)

INTERVENTIONS:
Drug: Apomorphine 0.25% (2.5mg/ml) — Apomorphine 0.5% (5mg/ml) will be diluted to 0.25% (2.5mg/ml) by the addition of the same volume physiological saline (NaCl 0.9%).
  Arms: Apomorphine 0.25% (2.5mg/ml)
Device: Massage with a spiky ball — Each patient will massage skin reactions with a spiky ball 3 times a day for 2 minutes.
  Arms: Massage with a spiky ball
Drug: Hydrocortisone cream 1% — Hydrocortisone cream 1% (1mg/g) will be administered on each nodule one time a day
  Arms: Hydrocortisone cream 1%
Drug: Subcutaneous hydrocortisone 10mg — Subcutaneous hydrocortisone 10mg will be administered previous to apomorphine infusion making use of the apomorphine infusion system
  Other Names: Solu-Cortef
  Arms: Subcutaneous hydrocortisone 10mg

SUMMARY:
Skin reactions as a result of continuous subcutaneous apomorphine infusion occur frequently and interfere with the absorption of apomorphine. The histopathology of apomorphine-induced skin reactions is poorly understood. Therefore treatment options are limited and suggestive.

Objective: to investigate the efficacy of four treatments including massage, dilution of apomorphine, treatment with topical hydrocortisone and pre-treatment with subcutaneous administered hydrocortisone, in Parkinson's disease patients with apomorphine-induced skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged ≥30;
* Diagnosis of idiopathic Parkinson's disease of >3 years' duration, defined by the United Kingdom (UK) Brain Bank criteria, with the exception of >1 affected relative being allowed, without any other known or suspected cause of Parkinsonism (Gibb & Lees, 1988);
* Treatment with continuous subcutaneous apomorphine infusion;
* Having apomorphine-induced skin reactions (i.e. erythema, swelling and/or nodule formation);
* Male and female patients must be compliant with a highly effective contraceptive method (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method) during the study, if sexually active;
* Subjects considered reliable and capable of adhering to the protocol, visit schedule, and medication intake according to the judgement of the investigator.

Exclusion Criteria:

* High suspicion of other parkinsonian syndromes;
* History of respiratory depression;
* Hypersensitivity to hydrocortisone or any excipients of the medicinal product;
* Concomitant therapy with histamine antagonist;
* Known with Cushing's disease or hypercortisolism
* Any medical condition that is likely to interfere with an adequate participation in the study including e.g. current diagnosis of unstable epilepsy; clinically relevant cardiac dysfunction and/or myocardial infarction or stroke within the last 12 months;
* Pregnant and breastfeeding women;
* Current infectious disease with fever at the time of investigation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes on global perceived effect scale | 14 days

SECONDARY OUTCOMES:
Changes in histological skin tissue characteristics | 14 days
  Histological skin tissue characteristics are presence of eosinophils, melanin-like pigment, fibrosis, lymphocytes and histiocytes.
Changes in nodule size (diameter) | 14 days
Changes in erythema size (diameter) | 14 days
Eosinophilia | 14 days
  Defined as increased absolute eosinophil count
Personal or family history of atopic constellation | 14 days
  Assessed with a questionnaire
Personal or family history of allergies | 14 days
  Assessed with a questionnaire

OTHER OUTCOMES:
Liver enzymes | 14 days
  aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), alkaline phosphatase (AF), lactate dehydrogenase (LDH), gamma-glutamyl transpeptidase (gGT)

CONTACTS AND LOCATIONS:
Overall Officials: Teus Van Laar, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Department of Neurology, Groningen, Netherlands

REFERENCES:
- [Derived] Borgemeester RWK, Diercks GFH, van Laar T. Treatment of subcutaneous nodules after infusion of apomorphine; a biopsy-controlled study comparing 4 frequently used therapies. Parkinsonism Relat Disord. 2021 Aug;89:38-40. doi: 10.1016/j.parkreldis.2021.06.024. Epub 2021 Jun 29. PMID 34218046